CLINICAL TRIAL: NCT05757141
Title: A Phase 1b/2 Open-label Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Exploratory Efficacy Following Fosigotifator Administration in Adult and Pediatric Subjects With Vanishing White Matter Disease
Brief Title: An Open-Label Exploratory Study of Fosigotifator in Participants With Vanishing White Matter Disease
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Calico Life Sciences LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: M23-523; 2023-505704-30-00 (Other: EU CT)
Record Dates: First submitted 2023-02-23; First posted 2023-03-07 (Actual); Last update posted 2025-11-12 (Actual); Status verified 2025-11

CONDITIONS: Vanishing White Matter Disease
Keywords: Neurodegenerative Diseases; Nervous System Diseases; Central Nervous System Brain Diseases; Hereditary Central Nervous System; Leukoencephalopathy with Vanishing White Matter
MeSH Terms: conditions — Leukoencephalopathies; Neurodegenerative Diseases; Nervous System Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (5):
- Fosigotifator - Cohort 1 (Experimental): Cohort 1: VWM adults >= 18 years.
  Interventions: Drug: Fosigotifator
- Fosigotifator - Cohort 1b (Experimental): Cohort 1b: VWM adults >= 18 years.
  Interventions: Drug: Fosigotifator
- Fosigotifator - Cohort 2 (Experimental): Cohort 2: VWM children>= 12 y and <18 years.
  Interventions: Drug: Fosigotifator
- Fosigotifator - Cohort 3 (Experimental): Cohort 3: VWM children >= 6 y and <12 years.
  Interventions: Drug: Fosigotifator
- Fosigotifator - Cohort 4 (Experimental): Cohort 4: VWM children >= 6 months and <6 years.
  Interventions: Drug: Fosigotifator

INTERVENTIONS:
Drug: Fosigotifator — Oral Use
  Other Names: ABBV-CLS-7262

SUMMARY:
Fosigotifator is an investigational drug being researched for the treatment of Vanishing White Matter disease in adult, pediatric and infant participants. This is a 201-week, open-label, multiple cohort study enrolling adults, pediatric and infant participants with Vanishing White Matter disease.

Participants will attend regular visits during the course of the study and complete medical assessments, blood tests, questionnaires, and be evaluated for side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females >= 6 months of age at the time of Screening.
2. Have VWM disease defined as:

   1. A clinical diagnosis by a physician experienced in the assessment of VWM disease; and
   2. A molecular diagnosis of VWM disease, and
   3. A magnetic resonance imaging (MRI) presentation consistent with VWM disease.
3. Have a designated caregiver who is able to complete the respective caregiver-centered assessments.
4. Signed and dated informed consent provided by the participant, or from a legally authorized representative (LAR) if participant is incapable to consent themselves.
5. Participants must meet criteria (a) and at least one of the following functional criteria (b or c):

   1. Medical history of at least 1 neurological symptom that is assessed by the investigator as having a reasonable possibility of being related to VWM disease.
   2. Motor criteria defined as inability to walk 10 or more steps with or without light support of 2 hands
   3. Cognitive criteria as assessed by the age-appropriate version of the Wechsler Intelligence Scale, with participants scoring < 50 on specific indices; specific details can be provided by the Study physician.
6. Pediatric participants in Cohort 4 must meet both criteria a and b below, or criterion c:

   1. Medical history of at least 1 neurological symptom that is assessed by the investigator as having a reasonable possibility of being related to VWM disease.
   2. Motor criteria as defined below:

   i. More than minimal head control as demonstrated by: While in prone position, the participant can lift his/her head and sustain the position for 10 seconds and bring his/her arms actively to weight bearing in that position.

   c. Presymptomatic and homozygous for Cree Leukoencephalopathy (EIF2B5 R195H) or other mutation with known imminent risk of significant clinical decline or death (sponsor must be notified and provide approval prior to screening and enrolling a participant that meets eligibility with only this criterion).
7. All male participants who are sexually active and not surgically sterilized must agree to use an acceptable contraceptive method. Additionally, male participants must agree to not donate sperm during the study until 30 days after the final dose of study drug.
8. All female participants who are sexually active and of childbearing potential must agree to use a highly effective contraceptive method. Additionally, female participants must agree to not donate eggs during the study and for 30 days after the final dose of study drug.

Exclusion Criteria:

1. Pediatric participants >= 6 months and < 6 years of age must not be on any form of respiratory support at the time of Screening.
2. Changes in medication use for the management of VWM disease symptoms within the 4 weeks preceding Screening.
3. Seizure disorder not considered adequately controlled by the investigator within the 6 months preceding Screening.
4. Participant who, in the opinion of the investigator, is incapable of completing study-required visits and procedures to assess primary and secondary endpoints.
5. Adult female participants who are pregnant, breastfeeding or providing breast milk.
6. Treatment with any other investigational treatment within 30 days or 5 half-lives (whichever is longer) prior to Baseline.
7. Any clinically significant laboratory or imaging findings at Screening.

Min Age: 6 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-03-13 (Actual); Primary Completion 2027-11 (Estimated); Study Completion 2029-11 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Baseline up to Approximately Day 28
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.03
Number of Participants with Change in Vital Signs | Baseline up to Approximately Day 28
  Number of Participants with Change in Vital Signs will be assessed.
Number of Participants with Change in ECG | Baseline up to Approximately Day 28
  Number of Participants with Change in ECG will be assessed.
Number of Participants with Change in Clinical Laboratory Tests | Baseline up to Approximately Day 28
  Number of participants with change in clinical laboratory tests will be assessed.
Change from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline up to Approximately Day 28
  The C-SSRS is a systematically administered instrument that reports the severity of both suicidal ideation and behavior, with a higher score denoting more severe suicidal ideation and behavior.
Plasma Concentration of Fosigotifator | Baseline up to approximately Week 96
  Maximum Plasma Concentration [Cmax]
Time to Cmax (Tmax) of Fosigotifator | Baseline up to approximately Week 96
  Tmax of Fosigotifator
Area Under the Plasma Concentration-Time Curve (AUC0-24h) of Fosigotifator | Baseline up to approximately Week 96
  AUC0-24h of Fosigotifator
Trough Concentration (Ctrough) of Fosigotifator | Baseline up to approximately Week 96
  Ctrough of Fosigotifator
Terminal Elimination Half-Life (t1/2) of Fosigotifator | Baseline up to approximately Week 96
  t1/2 of Fosigotifator

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | Baseline up to Approximately Week 197
  Number of patients with treatment-related adverse events as assessed by CTCAE v4.03
Number of Participants with Change in Vital Signs | Baseline up to approximately Week 197
  Number of Participants with Change in Vital Signs will be assessed.
Number of Participants with Change in ECG | Baseline up to approximately Week 197
  Number of Participants with Change in ECG will be assessed.
Number of Participants with Change in Clinical Laboratory Tests | Baseline up to approximately Week 197
  Number of participants with change in clinical laboratory tests will be assessed.
Change from Baseline in Columbia-Suicide Severity Rating Scale (C-SSRS) | Baseline up to approximately Week 197
  The C-SSRS is a systematically administered instrument that reports the severity of both suicidal ideation and behavior, with a higher score denoting more severe suicidal ideation and behavior.
Number of Participants with Change in Magnetic Resonance Imaging (MRI) | Baseline up to approximately Week 192
  Change in Brain Magnetic Resonance Imaging (MRI) associated with adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (5):
- United States (3):
  - Massachusetts General Hospital /ID# 270960, Boston, Massachusetts
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - University of Utah /ID# 255624, Salt Lake City, Utah
- McGill University Health Centre - Glen Site, Montreal, Quebec, Canada
- Amsterdam UMC, locatie VUmc /ID# 270955, Amsterdam, North Holland, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP
Time Frame: For details on when studies are available for sharing, visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M23-523